CLINICAL TRIAL: NCT00381563
Title: Bracing in Patellofemoral Osteoarthritis: A Clinical Trial
Brief Title: Knee Bracing for People With Patellofemoral Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-25641; P60AR047785 (NIH); 2P60AR047785-06 (NIH)
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Knee Osteoarthritis
Keywords: Bracing; Patellofemoral; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention to placebo (Other): Participants will wear the patellofemoral realigning knee brace for 6 weeks, followed by the non-aligning knee brace for 6 weeks.
  Interventions: Device: Patellofemoral realigning knee brace; Device: Non-aligning knee brace
- Placebo to intervetion (Other): Participants will wear the non-aligning knee brace for 6 weeks, followed by the patellofemoral realigning knee brace for 6 weeks.
  Interventions: Device: Patellofemoral realigning knee brace; Device: Non-aligning knee brace

INTERVENTIONS:
Device: Patellofemoral realigning knee brace — Knee brace that changes the tracking of the patella over the femur bone
Device: Non-aligning knee brace — Knee brace that does not change the tracking of the patella over the femur bone

SUMMARY:
Osteoarthritis, sometimes called degenerative joint disease, is the most common form of arthritis. It occurs when the cartilage in joints wears down over time. Symptoms can include pain, tenderness, stiffness, and inflammation. Studies have suggested that symptoms of knee osteoarthritis may be caused by abnormalities at the patellofemoral joint, which is the joint between the kneecap, called the patella, and the thigh bone, called the femur. This study will determine whether wearing a knee brace that realigns the patella over the femur is effective in relieving pain and improving function in adults with knee osteoarthritis.

DETAILED DESCRIPTION:
Bending and straightening at the knee causes the patella to glide along a groove in the femur bone. However, biomechanical imbalances can cause the patella to jump off track, which can lead to pain. Interventions that alter the load distribution across the patellofemoral joint, such as patella taping, may be helpful in alleviating symptoms. Patellar taping has in fact been shown to be effective in the short-term for treating patellofemoral osteoarthritis. But it has not been widely adopted in the clinical setting because it is complicated to administer, difficult to educate the patient about ongoing application, and lacks evidence of long-term efficacy. Also, patients often experience skin irritation from the taping and discomfort when removing the taping. An alternative treatment option is the use of a knee brace that realigns the tracking of the patella. This study will determine whether wearing a patellofemoral realigning knee brace is effective in relieving pain and improving function in adults with knee osteoarthritis.

Participation in this study will last about 3 to 9 months. All eligible participants will wear the same knee brace for a 2-week run-in period during which they will record when they wear the brace and any pain medication used. Next, participants will be randomly assigned to wear one of two knee braces for 6 weeks and a minimum of 4 hours each day. This will be followed by 6 weeks of wearing no knee brace, and then by 6 weeks of wearing whichever knee brace they did not wear during the first 6-week period. There will be a total of nine study visits. The first study visit will screen for eligible participants and will include an interview, knee evaluations, x-rays, and a urine pregnancy test. The second and sixth study visits will include knee evaluations, brace fittings, and instructions on how to correctly wear and adjust the brace. Most of the other study visits will consist primarily of interviews and functional tests. During the first and third 6-week periods, participants will maintain a log to record how long they wear their braces and any pain medication used. Participants will also wear an accelerometer, which will keep track of how many steps they take.

Participants will have the option of continuing in a 6-month follow-up period during which they can wear the brace of their choice. There will be three evaluations that will include questions on how participants are doing with their braces.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain on most days
* Either isolated patellofemoral osteoarthritis or mixed patellofemoral and tibiofemoral osteoarthritis, as based on x-ray

Exclusion Criteria:

* Bed- or chair-bound, usually uses an ambulation aid to walk (e.g., cane, crutch, or walker), or uses a wheelchair
* Pain emanating more from the back or hip than from the knee, as determined by screening questionnaire
* Low pain score on the visual analog scale (VAS) (less than 4 out of 10)
* Plans to move from the area within 10 months of study screening
* Symptomatic comorbid disease that limits activities more than knee pain does, as determined by screening questionnaire (e.g., congestive heart failure, chronic obstructive pulmonary disease)
* Receiving corticosteroid injections in the month before study entry, or receiving hyaluronan in the 6-month period before study entry. No other treatments will result in exclusion, although for patients taking glucosamine and/or chondroitin and/or a non-steroidal anti-inflammatory drug (NSAID), they must have taken these treatments for at least 2 months before study entry and must commit to not start a new treatment during the study.
* Bilateral total knee replacements or plans for a total knee replacement of the affected knee in the next 6 months
* Morbidly obese (body mass index greater than 35), as brace fitting and prevention of slippage of the brace will be difficult
* Known other causes of arthritis, including rheumatoid arthritis, systemic lupus erythematosus, gout, psoriatic arthritis, and pseudogout
* Skin breakdown at the site where the brace will be applied
* Failure to pass the run-in test, or the brace falls down the leg during the run-in

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hunter, MD, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Boston University, School of Medicine, Boston, Massachusetts
  - New England Baptist Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hunter DJ, Harvey W, Gross KD, Felson D, McCree P, Li L, Hirko K, Zhang B, Bennell K. A randomized trial of patellofemoral bracing for treatment of patellofemoral osteoarthritis. Osteoarthritis Cartilage. 2011 Jul;19(7):792-800. doi: 10.1016/j.joca.2010.12.010. Epub 2011 Jan 11. PMID 21232620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited through: public media including the Boston Metro, Community News, Baystate Banner and Tab, Craigslist; patients referred from BMC rheumatology, primary care, physical therapy, and orthopedics & from Baptist Hospital orthopedic clinics, and persons already recruited from studies whose consent forms allow contact
Groups:
- Placebo to Intervention: Participants will wear the non-aligning knee brace for 6 weeks, followed by the patellofemoral realigning knee brace for 6 weeks.
Period: Overall Study
Arm/Group | Intervention to Placebo | Placebo to Intervention
Started | 41 | 39
Completed | 34 | 33
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention to Placebo | Placebo to Intervention | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 53
  >=65 years | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.7) | 61 (9.1) | 60.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 41 | 39 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain on the VIsual Analog Scale (VAS)
Description: The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations, including those with rheumatic diseases. It is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (best) to the right (worst).The visual analog scale (VAS) pain ranges from 0-100
Time Frame: 6 weeks
Population: In this cross-over design where in one arm participants received the neutral brace with a realigning strap for the first 6 weeks then the neutral brace without a realigning strap for the second 6 weeks and the other arm used them in the opposite order, all 67 participants who completed the trial are re-grouped into the "intervention brace" group.
Measure: Mean (95% Confidence Interval); unit: change in units on a scale from baseline
Groups:
- Intervention Brace: All participants who completed the trial (n=67) are re-grouped into the "intervention brace" group.
Arm/Group | Intervention Brace
Number analyzed (Participants) | 67
change in units on a scale from baseline | -.068 [-6.2 to 4.8]

2. Primary Outcome: Change in WOMAC Pain Scale
Description: The WOMAC (Western Ontario and McMaster Osteoarthritis Index) is a widely used self-administered health status measure used in assessing pain, stiffness, and function in patients with OA of the hip or knee. It measures Pain (5 questions), Stiffness (2 questions), and Function (17 questions). The WOMAC pain scale ranges from 0-20. All the items are scored on a scale of 0-4 (0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely). Lower scores indicate lower levels of pain.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale change from baseline
Arm/Group | Intervention Brace
Number analyzed (Participants) | 67
units on a scale change from baseline | -0.11 [-0.66 to 0.88]

3. Secondary Outcome: Change in WOMAC Function Scale
Description: The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a self-administered health status measure for pain, stiffness, and function in patients with knee or hip OA. It measures Pain (5 questions), Stiffness (2 questions), and Function (17 questions). The WOMAC function score ranges from 0-68, all items are scored on a scale of 0-4 (0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely) for difficulty of specific functions. Lower overall function scores indicate higher levels of functioning or less difficulty performing a list of 17 specific activities.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale change from baseline
Arm/Group | Intervention Brace
Number analyzed (Participants) | 67
units on a scale change from baseline | -0.02 [-2.83 to 2.79]

ADVERSE EVENTS:
Arm/Group | Intervention to Placebo | Placebo to Intervention
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39

LIMITATIONS AND CAVEATS:
There was no control group without a brace for comparison to the intervention because of concerns about unblinding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No